CLINICAL TRIAL: NCT05379296
Title: Healthy Hearts: Leveraging the Diabetes Prevention Program to Decrease Health Disparities in Women of Reproductive Age
Acronym: HH
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Inadequate resources to complete within the required timeline.
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21-0325
Record Dates: First submitted 2022-05-02; First posted 2022-05-18 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2023-01

CONDITIONS: Prediabetic State; Gestational Weight Gain; Hypertension; Overweight or Obesity
Keywords: Prediabetic State; Gestational Weight Gain; Hypertension; Overweight or Obesity; Women's Health; Cardiovascular disease
MeSH Terms: conditions — Prediabetic State; Gestational Weight Gain; Hypertension; Overweight; Obesity; Cardiovascular Diseases | interventions — dentin sialophosphoprotein

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diabetes Prevention Program (DPP) (Active Comparator): CDC-approved 12-month DPP virtual lifestyle program
  Interventions: Behavioral: Diabetes Prevention Program (DPP)
- Diabetes Prevention Program Plus (DPP+) (Experimental): CDC-approved 12-month DPP virtual lifestyle program expanded to include a CDC-approved module on hypertension prevention and treatment
  Interventions: Behavioral: Diabetes Prevention Program Plus (DPP+)

INTERVENTIONS:
Behavioral: Diabetes Prevention Program Plus (DPP+) — The DPP+ includes the CDC-approved DPP lifestyle program expanded to include a CDC-approved module on hypertension prevention and treatment
  Arms: Diabetes Prevention Program Plus (DPP+)
Behavioral: Diabetes Prevention Program (DPP) — CDC-approved DPP lifestyle program
  Arms: Diabetes Prevention Program (DPP)

SUMMARY:
Nearly half of women have obesity and/or hypertension (HTN). Specific to women, pregnancy creates a vulnerable window for excess gestational weight gain (GWG), exacerbating intergenerational risks for obesity, HTN, type 2 diabetes (T2D), and cardiovascular disease (CVD) across the lifespan. Healthy lifestyles are the first-line recommendations for prevention and treatment of overweight/obesity, HTN, T2D, and CVD. The Diabetes Prevention Program (DPP) is a well-established, Centers for Disease Control and Prevention (CDC)-led public health program focusing on healthy lifestyle changes and is effective at reducing 5-7% of body weight, lowering risks for T2D. Interestingly, research investigating the DPP as a lifestyle intervention for other chronic conditions (i.e., overweight/obesity and HTN) is lacking, demonstrating a missed opportunity. The aim of this study is to determine the initial effects of the first 6-months and after receiving the full 12-months of the virtual DPP compared to the DPP expanded with a CDC-approved HTN prevention component (DPP+) on physical activity, diet, weight, and CVD risk factors in 30 prediabetic women (18-45 years old) with a history of excess GWG, overweight/obesity, and HTN. Participants will be recruited through University of Texas Medical Branch (UTMB) community-based clinics using Epic. The Participants will be randomized into 2 groups (DPP and DPP+) and guided through the 12-month virtual DPP or DPP+ program using UTMB DPP personnel.

ELIGIBILITY:
Inclusion Criteria:

* Women with prediabetes and eligible for the DPP, overweight/obesity, HTN (diagnosed or 3 successive high blood pressure readings), and history of excess gestational weight gain during most recent pregnancy

Exclusion Criteria:

* Pregnant and lactating women, participants planning to move out of Galveston County within the next year

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-01-20 (Estimated); Study Completion 2023-01-20 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Systolic Blood Pressure at 6 months | Baseline, 6-months
Change from Baseline Systolic Blood Pressure at 12 months | Baseline, 12-months
Change from Baseline Diastolic Blood Pressure at 6 months | Baseline, 6-months
Change from Baseline Diastolic Blood Pressure at 12 months | Baseline, 12-months
Change from Baseline High-density lipoproteins at 6 months | Baseline, 6-months
Change from Baseline High-density lipoproteins at 12 months | Baseline, 12-months
Change from Baseline Low-density lipoproteins at 6 months | Baseline, 6-months
Change from Baseline Low-density lipoproteins at 12 months | Baseline, 12-months
Change from Baseline Triglycerides at 6 months | Baseline, 6-months
Change from Baseline Triglycerides at 12 months | Baseline, 12-months
Change from Baseline Total cholesterol at 6 months | Baseline, 6-months
Change from Baseline Total cholesterol at 12 months | Baseline, 12-months
Change from Baseline Hemoglobin a1c at 6 months | Baseline, 6-months
Change from Baseline Hemoglobin a1c at 12 months | Baseline, 12-months
Change from Baseline Weight at 6 months | Baseline, 6-months
Change from Baseline Weight at 12 months | Baseline, 12-months
Change from Baseline Body mass index at 6 months | Baseline, 6-months
Change from Baseline Body mass index at 12 months | Baseline, 12-months
Change from Baseline Fasting blood glucose at 6 months | Baseline, 6-months
Change from Baseline Fasting blood glucose at 12 months | Baseline, 12-months
Change from Baseline Serum insulin at 6 months | Baseline, 6-months
Change from Baseline Serum insulin at 12 months | Baseline, 12-months

SECONDARY OUTCOMES:
Change from Baseline Total portions of Combined Weekly Fruit and Vegetable Consumption at 6 months | Baseline, 6-months
  Measured using the PreventT2 Diabetes Prevention Program questionnaire
Change from Baseline Total portions of Combined Weekly Fruit and Vegetable Consumption at 12 months | Baseline, 12-months
  Measured using the PreventT2 Diabetes Prevention Program questionnaire
Change from Baseline Total portions of Fried Food Consumption at 6 months | Baseline, 6-months
  Measured using the PreventT2 Diabetes Prevention Program questionnaire
Change from Baseline Total portions of Fried Food Consumption at 12 months | Baseline, 12-months
  Measured using the PreventT2 Diabetes Prevention Program questionnaire
Change from Baseline Objective Total Weekly Physical activity minutes at 6 months | Baseline, 6-months
  Measured using Fitbit Inspire 2
Change from Baseline Objective Total Weekly Physical activity minutes at 12 months | Baseline, 12-months
  Measured using Fitbit Inspire 2
Change from Baseline Subjective Weekly Physical activity at 6 months | Baseline, 6-months
  Stanford Brief Leisure-Time Activity Categorical Item (L-CAT 2.2)
Change from Baseline Subjective Weekly Physical activity at 12 months | Baseline, 12-months
  Stanford Brief Leisure-Time Activity Categorical Item (L-CAT 2.2)
Change from Baseline Visceral adiposity tissue at 6 months | Baseline, 6-months
  Measured using Dual energy X-ray absorptiometry
Change from Baseline Visceral adiposity tissue at 12 months | Baseline, 12-months
  Measured using Dual energy X-ray absorptiometry
Change from Baseline C-reactive protein at 6 months | Baseline, 6-months
Change from Baseline C-reactive protein at 12 months | Baseline, 12-months

CONTACTS AND LOCATIONS:
Overall Officials: Crystal Clark Douglas, PhD, Principal Investigator — University of Texas

IPD SHARING:
Plan to Share IPD: No